CLINICAL TRIAL: NCT04087421
Title: Comparison of Transanal Irrigation and Glycerol Suppositories in Treatment of Low Anterior Resection Syndrome: A Multicentre Randomised Controlled Trial
Brief Title: Comparison of Transanal Irrigation and Glycerol Suppositories in Treatment of Low Anterior Resection Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 676869
Record Dates: First submitted 2019-08-26; First posted 2019-09-12 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-02

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
Keywords: Low Anterior Resection Syndrome; Transanal irrigation; Glycerol suppositories
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transanal irrigation (Experimental): Participants receiving TAI will irrigate once/day with stepwise volumes; 1. month 150 ml, 2. month 300 ml, and 3. month 500 ml.
  Interventions: Device: Qufora Irrisedo Cone System
- Glycerol suppositories (Active Comparator): Participants treated with glycerol suppositories will administer one glycerol suppository once/day.
  Interventions: Drug: Glycerol "OBA"

INTERVENTIONS:
Device: Qufora Irrisedo Cone System — The system works by connecting a tube from a water bag to a cone. The cone is placed into the rectum and the prescribed water volume is pumped into the rectum. When the water has been installed the valve is closed and the cone removed. Residual water and stool will then flow into the toilet.
  Arms: Transanal irrigation
Drug: Glycerol "OBA" — Rectal suppository. Stimulates the rectum and softens and loosens stool.
  Arms: Glycerol suppositories

SUMMARY:
The study is a multicentre randomized controlled trial with the objective to compare the effect of transanal irrigation with glycerol suppositories in patients suffering from major Low Anterior Resection Syndrome (LARS).

DETAILED DESCRIPTION:
Transanal irrigation (TAI) is used as a second-line treatment following unsuccessful personalised conservative treatment (PCT) of LARS. However, it is unknown if scheduled, initiated defecation with the aid of a glycerol suppository will have the same clinical effect as TAI. Thus, the aim of this study is to compare the effect of TAI with a glycerol suppository in patients suffering from major LARS.

The study is a multi-centre, randomised, controlled, 12 weeks, parallel-group trial comparing treatment with TAI to treatment with glycerol suppositories. Patients will be randomised - stratified by centre and neoadjuvant radiotherapy - in a 1:1 ratio to receive treatment with TAI or glycerol suppositories. Primary endpoint will be assessed by the end of week twelve.

ELIGIBILITY:
Inclusion Criteria:

* Patients electively treated for rectal cancer with a low anterior resection.
* Unsuccessful PCT after at least 4 weeks of treatment for LARS (LARS score >29 at evaluation).
* At least 3 months after surgery (including reversal of a temporary loop-ileostomy).
* Age >= 18 years
* Ability to understand written and spoken language actual for the including site (due to questionnaire validity).

Exclusion Criteria:

* Former use of TAI
* Prior systematic use of rectal emptying aids
* Anastomotic stenosis
* History of anastomotic leakage
* Current metastatic disease or local recurrence
* Ongoing oncological treatment
* Postoperative radiotherapy for rectal cancer
* Previous or current cancer in other pelvic organs than the rectum
* Underlying diarrhoeal disease
* Inflammatory bowel disease
* Dementia
* Spinal cord injury, multiple sclerosis, Parkinson's disease or other significant neurologic disease assessed to be a contributory cause to LARS symptoms.
* Inability of patient to use TAI
* Inability and unwillingness to give informed consent
* Pregnancy or intention to become pregnant during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bowel function, change in symptom 1 score assessed using the Measure Yourself Medical Outcome Profile (MYMOP2) Score. | 12 weeks.
  MYMOP2 is a validated problem-specific, patient-generated questionnaire. Patients are asked to specify one or two symptoms that concern them the most. Subsequently they evaluate the severity on a 7-point Likert scale. The second part of the questionnaire uses the same scale to assess whether the symptom limits or prevent any daily activity, and also to rate general well-being. Follow-up questionnaires address the original issues completed in the initial form. Symptom 1, symptom 2, activity, and wellbeing each have a separate score between 0 and 6 with 0 indicating "as good as it could be" and 6 "as bad as it could be". An overall score is calculated by taking the average of item scores.

SECONDARY OUTCOMES:
Bowel function, change in symptom 2 score assessed using the Measure Yourself Medical Outcome Profile (MYMOP2) Score. | 4, 8, and 12 weeks.
  MYMOP2 is a validated problem-specific, patient-generated questionnaire. Patients are asked to specify one or two symptoms that concern them the most. Subsequently they evaluate the severity on a 7-point Likert scale. The second part of the questionnaire uses the same scale to assess whether the symptom limits or prevent any daily activity, and also to rate general well-being. Follow-up questionnaires address the original issues completed in the initial form. Symptom 1, symptom 2, activity, and wellbeing each have a separate score between 0 and 6 with 0 indicating "as good as it could be" and 6 "as bad as it could be". An overall score is calculated by taking the average of item scores.
Change in activity score assessed using the Measure Yourself Medical Outcome Profile (MYMOP2) Score. | 4, 8, and 12 weeks.
  MYMOP2 is a validated problem-specific, patient-generated questionnaire. Patients are asked to specify one or two symptoms that concern them the most. Subsequently they evaluate the severity on a 7-point Likert scale. The second part of the questionnaire uses the same scale to assess whether the symptom limits or prevent any daily activity, and also to rate general well-being. Follow-up questionnaires address the original issues completed in the initial form. Symptom 1, symptom 2, activity, and wellbeing each have a separate score between 0 and 6 with 0 indicating "as good as it could be" and 6 "as bad as it could be". An overall score is calculated by taking the average of item scores.
Change in well-being score assessed using the Measure Yourself Medical Outcome Profile (MYMOP2) Score. | 4, 8, and 12 weeks.
  MYMOP2 is a validated problem-specific, patient-generated questionnaire. Patients are asked to specify one or two symptoms that concern them the most. Subsequently they evaluate the severity on a 7-point Likert scale. The second part of the questionnaire uses the same scale to assess whether the symptom limits or prevent any daily activity, and also to rate general well-being. Follow-up questionnaires address the original issues completed in the initial form. Symptom 1, symptom 2, activity, and wellbeing each have a separate score between 0 and 6 with 0 indicating "as good as it could be" and 6 "as bad as it could be". An overall score is calculated by taking the average of item scores.
Bowel function assessed using the Low Anterior Resection Syndrome (LARS) Score. | 4, 8, and 12 weeks.
  The LARS score is a validated questionnaire for evaluation of bowel function after sphincter-preserving surgery. It covers five LARS symptoms including: incontinence for flatus, incontinence for liquid stools, frequency (number of daily bowel movements), clustering, and urgency. The scores from each five answers are added to one final score. The score ranges from 0-42 with 0 indicating the best score and 42 the worst. Based on the score patients are stratified into: 0-20: No LARS, 21-29: Minor LARS, 30-42: Major LARS.
Bowel function assessed using the Memorial Sloan-Kettering Cancer Centre Bowel Function Instrument (MSKCC BFI) Score. | 4, 8, and 12 weeks.
  The MSKCC BFI score is a validated questionnaire for evaluation of bowel function after sphincter-preserving surgery. It comprises 18 items covering the frequency of various LARS symptoms and is divided into three sub-scales and four single items. It is scored on a 5-point Likert scale ranging from "always" to "never". The sub-scales scores are summarised as: A 6-item frequency sub-scale (6-30), a four-item dietary sub-scale (4-20), and a four-item urgency sub-scale (4-20). A global score can be calculated as the sum of the sub-scale scores. A total score (possible score range 18-90) can be calculated by adding all the item scores (sub-scale scores plus single item scores). A higher score indicates better bowel function.
Frequency of bowel movements, incontinence episodes (total, passive, and urge), urge episodes, soiling, and daily gas incontinence, incomplete emptying, and average urge time assessed using the Journl A/S application. | Weeks 3-4, weeks 7-8, and weeks 11-12.
  Journl A/S has developed an application for evaluation of bowel function. The participants can enter real-time data into the application and data will be stored in a backend allowing calculations of frequencies and averages on these parameters during weeks 3-4, 6-8, and 11-12 in the study period.
Fecal incontinence assessed using the St. Mark's Incontinence Score. | 4, 8, and 12 weeks.
  The St. Mark's Incontinence score is a validated questionnaire for evaluation of fecal incontinence. It covers the frequency of three types of fecal incontinence: Solid, liquid, and gas and the consequences: Pad wearing or usage of a plug, and lifestyle alteration. Furthermore, it incorporates: urgency and the need for antidiarrheal drugs. For each item of fecal incontinence and lifestyle alterations the frequency option ranges from never (score 0) to daily (score 4). The rest of the items are scored as follows: Urgency: No (score 0) or yes (score 4), antidiarrheal drugs: No (score 0) or yes (score 2), pad wearing: No (score 0) or yes (score 2). The total score is the sum of each item. The minimum score is 0 = no incontinence and maximum score is 24 = totally incontinent.
Female urinary function assessed using the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS). | 12 weeks.
  The ICIQ-FLUTS questionnaire is validated for evaluating female lower urinary tract symptoms. It consists of 12 items which are all scores from 0-4 and the overall score ranges from 0-48. A higher score indicates a worse condition. A filling sub-scale (0-16), a voiding sub-scale (0-12), and an incontinence symptoms sub-scale can be calculated (0-20).
Male urinary function assessed using the International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms (ICIQ-MLUTS). | 12 weeks.
  The ICIQ-MLUTS questionnaire is validated for evaluating male lower urinary tract symptoms. It consists of 13 items which are all scores from 0-4 and the overall score ranges from 0-52. A higher score indicates a worse condition. A voiding sub-scale (0-20) and an incontinence symptoms sub-scale (0-24) can be calculated.
Female sexual function assessed using The Rectal Cancer Female Sexuality Score. | 12 weeks.
  The Rectal Cancer Female Sexuality Score is a validated questionnaire for assessment of sexuality after treatment for rectal cancer. The score includes 7 items and ranges from 0-29. A score >= 9 indicates sexual dysfunction.
Male sexual function assessed using the 5-item International Index of Erectile Function (IIEF-5). | 12 weeks.
  The 5-item International Index of Erectile Function (IIEF-5) Questionnaire is a 5-question validated questionnaire for assessment of erectile dysfunction (ED). The possible scores range from 5-25 and the severity of ED is classified into five categories stratified by score: 22-25 (no ED), 17-21 (mild), 12-16 (mild to moderate), 8-11(moderate), 5-7 (severe).
Quality of life assessed using the EORTC Quality of Life questionnaire (QLQ)-C30. | 12 weeks.
  The European Organisation for Research and Treatment of Cancer (EORTC) developed and validated a 30-item core questionnaire (QLQ-C30) reflecting global QoL in cancer patients. QLQ-C30 comprises five functional scales, three symptom scales, a global health scale/ a quality of life scale, and six single items. All the scales and single item measures range in score from 0-100. A high score represents a higher level of functioning, a high quality of life, and a greater degree of symptoms.
Quality of life assessed using the EORTC Quality of Life questionnaire (QLQ)-CR29. | 12 weeks.
  QLQ-CR29 is developed by The European Organisation for Research and Treatment of Cancer (EORTC). It is a validated supplement to the QLQ-C30 specifically designed for assessment of quality of life in colorectal cancer patients. QLQ-CR29 consists of four functional scales and eighteen single items. All the scales range from 0-100. A high score represents a higher level of functioning and a greater degree of symptoms.
Impact on quality of life and activities assessed using the Journl A/S application. | Weeks 3-4, weeks 7-8, and weeks 11-12.
  Journl A/S has developed an application for evaluation of bowel function and impact on quality of life and activity. The participants can enter real-time data into the application and data will be stored in a backend allowing daily evaluation of quality of life and activity during weeks 3-4, 6-8, and 11-12 in the study period.
Quality of life and Health economics assessed using the European Quality of Life-5 Dimensions 5-level version questionnaire (EQ-5D-5L). | 12 weeks.
  The EQ-5D-5L is a standardised measure of health status developed by the EuroQoL Group. It consists of a descriptive system and a EQ Visual Analogue scale. Each dimension in the descriptive system has five levels: No problems, slight problems, moderate problems, severe problems, and extreme problems. Each dimension is referred to in terms of a 5-digit code. The EQ Visual Analogue scale records the respondent's self-rated health on a vertical scale ranging from 0-100 where the endpoints are labelled "best imaginable" (100) and "worst imaginable" (0). The EQ-5D-5L can be converted into an index value which facilitates the calculation of quality-adjusted life years (QALYs) that are used in economic evaluations of health care interventions.
Health economics assessed using the ICEpop CAPability measure for Adults (ICECAP-A). | 12 weeks.
  The ICECAP-5 is a validated questionnaire for measure of capability for the general adult population for use in economic evaluation. It covers: attachment, stability, achievement, enjoyment, and autonomy. Each item is scored from 1-4 with 4 indicating the best capability and 1 the worst. A total score can be calculated ranging from 5-20. Furthermore, a weighted score can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, Principal Investigator — Research Unit, Dept. of Surgery, Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Department of Surgery, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No